CLINICAL TRIAL: NCT07309081
Title: Effect of Soleus Muscle Kinetic Control Training on Gait and Electromyographic Activity in Patients With Stroke
Acronym: EMG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Habiba Mohamed Ahmed Mahmoud, principle investigator : habiba mohamed ahmed mahmoud, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/006089
Record Dates: First submitted 2025-12-01; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: kinetic control; gait; EMG; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: kinetic and traditional therapy
Who Masked: Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- soleus kinetic control (Experimental): twenty patients will receive soleus kinetic control plus conventional physiotherapy three times a week for 8 weeks
  Interventions: Other: soleus kinetic control; Other: conventional therapy
- conventional therapy (Active Comparator): twenty patients will receive conventional physiotherapy three times a week for 8 weeks
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: soleus kinetic control — patients will receive kinetic control for 30 minutes structural progressive training for the soleus muscle guided by the EMG biofeedback plus conventional therapy; 1)Start in crook lying position with the heels level with the pelvis and lift the pelvis clear of the floor followed by bilateral heel raise,2)Progress further by shifting weight onto one leg and holding the heel raise and slowly lowering eccentrically on 1 foot, the next progression is to perform the same movement with the heels lower than the pelvis on step -below the pelvis. The exercise graduation will be guided by the visual EMG Biofeedback participants will receive feedback on soleus activation throughout the training.
  Arms: soleus kinetic control
Other: conventional therapy — the patients will receives conventional physiotherapy program static stretching and stretching board for calf muscle, stretching board, and push off exercises by having the patient push against the therapist or a treatment table during forward gait ( 30 minute), static stretch(30sec\set , rest 20sec\set total 5 set, 3 times \week , for 8 week ), stretching board (4 min\set , rest 1 min\set total 2 set , 3 times \week , for 8 week ) (10 minute) push off training (15 minute 3 times \week , for 8 week )x2

SUMMARY:
this study was designed to investigate the effect of soleus muscle kinetic control training on Gait and electromyographic activity of the calf muscle in patients with stroke

DETAILED DESCRIPTION:
Stroke is a neurological condition characterized by a reduced blood supply to the brain tissue, resulting in paralysis of part or all of the body, limiting physical activity and social participation. Gait impairment accounts for the largest proportion of physical activity limitations in stroke patients and is characterized by muscle weakness, foot drop, spasticity, and foot deformity .Gait abnormalities following stroke are often disabling. Reduced ankle dorsiflexion, knee flexion, or hip flexion torques are often postulated causes of compromised toe clearing during the swing phase of gait. conversely, gait asymmetry and reduced walking speed has been attributed to weakness of the planter flexors.The kinetic control comprises balanced presentation of the movement choices with ideal interaction among the key components for the sensorimotor neuromuscular control that mediated by afferent sensory input, particularly the proprioceptive input, CNS integration, optimal motor co-ordination, and physiological stresses to assure functional dynamic stability and controlled mobility. forty patients with stroke will be assigned to two groups; one group will recieve kinetic control plus conventional therapy and control group will receive conventinoal therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or hemorrhagic stroke, as confirmed by CT and or MRI scan.
* Age of the patients between 45 to 60 years old.
* Ability to walk a minimum of 10 m with or without some physical assistance from a therapist (functional ambulation category more than 2).
* Demonstrate weakness of the foot muscles, measured by muscle function tests according Medical Research council scale more than 3.
* Muscle tone of the affected lower limb ranges from 1 to +1 according to modified Ashworth scale.

Exclusion Criteria:

* Unilateral neglect, hemianopia, or apraxia
* Having any other neurological disorder affecting their lower extremities e.g. MS, Parkinsonism, peripheral neuropathy.
* Patients with previous fractures in lower limb (Ankle or foot).
* Patients with musculoskeletal disorder such as severe arthritis, ankle surgery, leg length discrepancy or contractures of fixed deformity of ankle joint.
* Patients with visual, auditory impairment affecting their ability to complete tasks.
* Patients with cognitive impairments

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
muscle amplitude | up to eight weeks
  A steady device will be used to assess muscle amplitude in the form of RMS with microvolt as the measurement unit
giat function | up to eight weeks
  The Dynamic Gait Index (DGI) is an ordinal test of gait function evaluates the capacity to adapt gait to complex walking tasks encountered in everyday life. Eight aspects of gait are scored based on observation as the patient walks over a 6.1-m level surface.
  The rater records an ordinal score that ranges from 0 (unable or done very poorly) to 3 (normal score) for a total point value of 24. Scores of less than 21 appear to suggest risk for falls
Gait Cycle time | up to eight weeks
  time of gait cycle (seconds) will be measured by steady device
step time | up to eight weeks
  the time of step by seconds will be measured by steady device
cadence | up to eight weeks
  Cadence, number of steps per minute, will be measured by steady device
stance phase percentage | up to eight weeks
  the percentage of stance phase will be measured by steady device
swing phase percentage | up to eight weeks
  the percentage of swing phase will be measured by steady device
single and double support percentage | up to eight weeks
  single and double support percentage of gait cycle will be measured by steady device
first and second double support percentage | up to eight weeks
  first and second double support percentage of gait cycle will be measured by steady devcie
stride length | up to eight weeks
  stride length by cm will be measured by steady device
gait speed | up to eight weeks
  gait speed by km/h will measured by steady device